CLINICAL TRIAL: NCT04057144
Title: Acceptance and Commitment Therapy With and Without Enhanced Mindfulness Training for Chronic Pain: A Randomized Controlled Efficacy and Mediator Study
Brief Title: Acceptance and Commitment Therapy With and Without Enhanced Mindfulness Training for Chronic Pain
Acronym: MUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Oslo University Hospital (Other); University Hospital of North Norway (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/503
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
Keywords: Mindfulness; Psychotherapy, Group; Behavior Therapy
MeSH Terms: conditions — Chronic Pain | interventions — Sound Recordings; Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: This is a three group randomized controlled trial with 162 patient in each group, six different measurement points, of which pre-treatment and 52 weeks after start of the treatment are the crucial points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT with mindfulness (Experimental): 4-hour weekly session of acceptance and commitment therapy (ACT) with mindfulness exercises during 8 weeks in groups of 8
  Interventions: Behavioral: ACT; Behavioral: mindfulness exercises and audio recordings
- ACT without mindfulness (Experimental): 4-hour weekly acceptance and commitment therapy (ACT) without mindfulness exercises during 8 weeks in groups of 8
  Interventions: Behavioral: ACT
- Education program (Active Comparator): Self-management education program during 8 weeks in groups of 8.
  Interventions: Behavioral: Education program

INTERVENTIONS:
Behavioral: ACT — Acceptance and commitment therapy (ACT) sessions, lead by 2 qualified therapists, using a manual based on Steven Hayes et al 1999 that was adapted to group therapy and includes all the dynamic processes of ACT.
  Arms: ACT with mindfulness; ACT without mindfulness
Behavioral: mindfulness exercises and audio recordings — mindfulness exercises introduced in the ACT sessions. In addition daily home meditation exercises based on the program developed by Kabat-Zinn 2005 and with help of audio recordings.
  Arms: ACT with mindfulness
Behavioral: Education program — Self-management education program. Information given by a qualified health professional on pain and symptom management, stress, sleep, eating habits, mental health problems. Group discussions about thoughts and experiences.
  communication skills and physical activity
  Arms: Education program

SUMMARY:
As non-pharmacological alternatives, psychosocial treatments have been recommended for chronic pain management. One such treatment is Acceptance and Commitment Therapy (ACT). ACT is a cognitive behavior therapy based on Relational Frame Theory, a comprehensive theory about language and cognition. This treatment intends to help patients identify values ("what is truly meaningful to them") and to set goals and take action according to their values. ACT has research support in the treatment of several mental health problems. Moreover patients are taught mindfulness skills to increase acceptance of pain, thoughts and feelings so that these will have less impact on functioning and action. Among patients with chronic pain, several small clinical trials have shown that ACT is more effective than other treatments in terms of increasing function and improving mental health. ACT in combination with mindfulness training has not been tested so far. Further methodologically robust trials are required. This study will therefore examine whether ACT is more effective for chronic pain than an education program, and whether adding daily mindfulness training will improve the outcome, in a large sample of patients from four multidisciplinary pain centers.

ELIGIBILITY:
Inclusion Criteria:

* referred to one of the pain clinics in Oslo (200), Trondheim (200), Bergen (100) or Tromsø (100)
* primary diagnosis of chronic pain lasting for at least 6 months

Exclusion Criteria:

* severe somatic disease
* severe mental disorder (ongoing mania, psychosis, suicidal ideation, substance abuse/addiction
* not able to communicate in Norwegian
* needing 24-hour personal assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
pain intensity measured by the Norwegian Brief Pain Inventory (BPI) | 44 weeks after end of treatment
  the Brief Pain Inventory includes four 0-10 numerical rating scales: for 'pain now', and for 'least pain', 'worst pain', and 'average pain' during the last 24 hours, with 0 = no pain to 10 = pain as bad as you can imagine. A pain severity index is calculated by adding the scores on the pain severity items

SECONDARY OUTCOMES:
pain intensity measured by the Norwegian Brief Pain Inventory (BPI) | 8 weeks after end of treatment
  the Brief Pain Inventory includes four 0-10 numerical rating scales: for 'pain now', and for 'least pain', 'worst pain', and 'average pain' during the last 24 hours, with 0 = no pain to 10 = pain as bad as you can imagine. A pain severity index is calculated by adding the scores on the pain severity items
pain intensity measured by the Norwegian Brief Pain Inventory (BPI) | 24 weeks after end of treatment
  the Brief Pain Inventory includes four 0-10 numerical rating scales: for 'pain now', and for 'least pain', 'worst pain', and 'average pain' during the last 24 hours, with 0 = no pain to 10 = pain as bad as you can imagine. A pain severity index is calculated by adding the scores on the pain severity items
pain intensity measured by the Norwegian Brief Pain Inventory (BPI) | 3 years after end of treatment
  the Brief Pain Inventory includes four 0-10 numerical rating scales: for 'pain now', and for 'least pain', 'worst pain', and 'average pain' during the last 24 hours, with 0 = no pain to 10 = pain as bad as you can imagine. A pain severity index is calculated by adding the scores on the pain severity items
physical function | 8 weeks after end of treatment
  according to the SF-36 Health Survey
physical function | 24 weeks after end of treatment
  according to the SF-36 Health Survey
physical function | 44 weeks after end of treatment
  according to the SF-36 Health Survey
physical function | 3 years after end of treatment
  according to the SF-36 Health Survey
mental health | 8 weeks after end of treatment
  according to the SF-36 Health Survey
mental health | 24 weeks after end of treatment
  according to the SF-36 Health Survey
mental health | 44 weeks after end of treatment
  according to the SF-36 Health Survey
mental health | 3 years after end of treatment
  according to the SF-36 Health Survey

OTHER OUTCOMES:
attentional functioning | 8 weeks after end of treatment
  assessed by the Attention Network Test (Fan et al 2002) specifically designed to measure alerting, orienting and executive attention within a single testing session, which can be reported from the patients computer and lasts about 15 min
attentional functioning | 24 weeks after end of treatment
  assessed by the Attention Network Test (Fan et al 2002) specifically designed to measure alerting, orienting and executive attention within a single testing session, which can be reported from the patients computer and lasts about 15 min
attentional functioning | 44 weeks after end of treatment
  assessed by the Attention Network Test (Fan et al 2002) specifically designed to measure alerting, orienting and executive attention within a single testing session, which can be reported from the patients computer and lasts about 15 min

CONTACTS AND LOCATIONS:
Overall Officials: Tormod Landmark, phd, Principal Investigator — St. Olavs Hospital
Locations (4):
- Norway (4):
  - Haukeland universitetssykehus, Bergen
  - Oslo universitetssykehus, Oslo
  - Norges arktiske universitet, Tromsø
  - St Olavs Hospital, Trondheim

REFERENCES:
- [Derived] Nost TH, Woodhouse A, Dale LO, Hara KW, Steinsbekk A. Participants' experiences from group-based treatment at multidisciplinary pain centres - a qualitative study. Scand J Pain. 2021 Aug 30;22(2):365-373. doi: 10.1515/sjpain-2021-0099. Print 2022 Apr 26. PMID 34453878

DOCUMENTS (2):
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT04057144/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT04057144/SAP_001.pdf